CLINICAL TRIAL: NCT02473458
Title: Efficacy of Whole Extract of Licorice in Neurological Improvement of Patients After Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Afshin Borhani-Haghighi, Associate professor of Neurology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 90-01-01-4806
Record Dates: First submitted 2015-05-30; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Acute Stroke
Keywords: Licorice; Glycyrrhizic acid; Ischemic Stroke; Acute
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): patients with acute ischemic stroke who received standard care plus placebo filled capsules,
  Interventions: Drug: Placebo
- 450 mg licorice (Experimental): patients with acute ischemic stroke who received standard care plus capsules filled with 450 mg of whole extract of licorice.
  Interventions: Drug: Licorice whole extract
- 900 mg licorice (Experimental): patients with acute ischemic stroke who received standard care plus capsules filled with 900 mg of whole extract of licorice.
  Interventions: Drug: Licorice whole extract

INTERVENTIONS:
Drug: Licorice whole extract — Patients randomly received one of below capsules labeled with codes during the first 24 hours after stroke attack:
  1. Starch-filled capsules (as placebo)
  2. 450 mg whole licorice extract capsules
  3. 900 mg whole licorice extract capsules
  Arms: 450 mg licorice; 900 mg licorice
Drug: Placebo
  Arms: Control

SUMMARY:
Stroke is one of the most important causes of mortality and disability both in developed and developing countries. The only food and drug administration (FDA) approved therapy for acute stroke is recombinant tissue plasminogen activator (rtPA). But narrow therapeutic window has limited the usefulness of thrombolytic therapy. Therefore, finding effective neuroprotective drugs for the patients for whom thrombolysis is contraindicated or not feasible seemed to be mandatory in the world of cerebrovascular medicine.

Licorice, extracted from root of a plant scientifically known as Glycyrrhiza glabra, is used in food industries. Certain medical properties has been contributed to licorice and specifically to its active chemical components such as flavonoids and glycyrrhizic acid (GA). GA has been revealed to assert its anti-inflammatory effect by suppression of NF-κB, a key component of lipopolysaccharide-induced inflammatory response. Neuroprotective characteristics of GA has been widely investigated in recent studies.

In the present study, the investigators verified the efficacy and safety of oral administration of two different doses licorice extract in the patients with acute ischemic stroke, in a double-blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of acute ischemic stroke
* ROSIER score higher than 2
* Confirmation of ischemic brain damage in CT scan

Exclusion Criteria:

* Clinically relevant preexisting neurological deficit or previous CVA
* Primary intracerebral hemorrhage
* Coma (level of consciousness more than 2 in NIHSS scale).
* Negative swallow test
* Patients undergoing hemicraniectomy
* History of epilepsy
* Clinical seizure at onset of stroke
* Systolic BP is >160 mmHg, diastolic BP>110 at onset of stroke (if a rise in blood pressure occurred in the course of study it was controlled according to medical guidelines)
* Atrial fibrillation or other tachy/bradyarrythmias at time of allocation or in the middle of intervention
* Ejection Fraction less than 45%
* Potassium less than 4 mEq/dl at onset of stroke
* Malignancy or premalignant state within 5 years
* Myocardial infarction in previous month
* Significant kidney disease (creatinine higher than 1.8 mg/dl)
* Significant liver disease (Bilirubin > 20 mmoll/L)
* Significant lung disease (FEV1 < 1.5 L, pO2 < 70 in room air, pCO2 > 45)
* Psychiatric illness requiring hospital admission
* Warfarin intake
* Digoxin intake
* Pregnancy
* Breast feeding
* Inability to have follow/up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of neurological status of the patient measured by National Institute of health stroke Scale (NIHSS) after hospital stay | Atfer hospital stay, 5-14 days
  This scale is a standard measurement of neurological status of the patient
Change from baseline of neurological status of the patient measured by Modified Rankin Scale after hospital stay | Atfer hospital stay, 5-14 days
  This scale is a standard measurement of neurological status of the patient
Change from baseline of neurological status of the patient measured by National Institute of health stroke Scale (NIHSS) after 3 months | 3 months after stroke
Change from baseline of neurological status of the patient measured by Modified Rankin Scale after 3 months | 3 months after stroke

SECONDARY OUTCOMES:
Blood sugar | Participants were followed during their hospital stay for an average duration of 5 days
  For measurement of possible hyperglycemic effect
Blood pressure | Participants were followed during their hospital stay for an average duration of 5 days
  For detection of possible of occurrence hypertension due to pseudo-hyperaldosteronism effect of licorice
Serum Na and K | Participants were followed during their hospital stay for an average duration of 5 days
  For detection of possible of occurrence hypertension due to pseudo-hyperaldosteronism effect of licorice

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Departement of Namazi hospital, Shiraz, Fars, Iran

REFERENCES:
- [Background] Hinkle JL, Guanci MM. Acute ischemic stroke review. J Neurosci Nurs. 2007 Oct;39(5):285-93, 310. doi: 10.1097/01376517-200710000-00005. PMID 17966295
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):e6-e245. doi: 10.1161/CIR.0b013e31828124ad. Epub 2012 Dec 12. No abstract available. PMID 23239837
- [Background] Granitto M, Galitz D. Update on stroke: the latest guidelines. Nurse Pract. 2008 Jan;33(1):39-46; quiz 47. doi: 10.1097/01.NPR.0000305977.24952.1c. No abstract available. PMID 18192863
- [Background] Ramos-Cabrer P, Campos F, Sobrino T, Castillo J. Targeting the ischemic penumbra. Stroke. 2011 Jan;42(1 Suppl):S7-11. doi: 10.1161/STROKEAHA.110.596684. Epub 2010 Dec 16. PMID 21164112
- [Background] Hwang IK, Lim SS, Choi KH, Yoo KY, Shin HK, Kim EJ, Yoon-Park JH, Kang TC, Kim YS, Kwon DY, Kim DW, Moon WK, Won MH. Neuroprotective effects of roasted licorice, not raw form, on neuronal injury in gerbil hippocampus after transient forebrain ischemia. Acta Pharmacol Sin. 2006 Aug;27(8):959-65. doi: 10.1111/j.1745-7254.2006.00346.x. PMID 16867245